CLINICAL TRIAL: NCT05614375
Title: Prospective Observational Single Arm Study of Endoscopic Surgery in the Treatment of Soft Tissue Sarcoma in Nasal and Paranasal Sinus
Brief Title: Endoscopic Surgery in the Treatment of Soft Tissue Sarcoma in Nasal and Paranasal Sinus
Status: Recruiting | Type: Observational
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: SNSTS-SA-01-V1
Record Dates: First submitted 2021-12-09; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Sarcoma,Soft Tissue; Nasal Cavity Cancer; Paranasal Sinus Cancer; Surgery
Keywords: soft tissue sarcoma; nasal cavity and paranasal sinus; endoscopic surgery; prognose; overall survival rate; outcome; quality of life
MeSH Terms: conditions — Sarcoma; Paranasal Sinus Neoplasms | interventions — Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — tumor，para-carcinoma tissue，venous blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- soft tissue sarcoma with endoscopic surgery: patients with soft tissue sarcoma accept endoscopic surgery
  Interventions: Procedure: endoscopic surgery

INTERVENTIONS:
Procedure: endoscopic surgery — transnasal endoscopic surgery

SUMMARY:
Soft tissue sarcoma (STS) refers to a group of malignant tumors derived from non-epithelial extraosseous tissues, mainly from the mesoderm, partly from the neuroectoderm, including muscle, fat, fibrous tissue, blood vessels and peripheral nerves . STS is divided into 12 major categories based on tissue origin. According to different morphologies and biological behaviors, there are more than 50 subtypes. The most common subtypes include: undifferentiated pleomorphic sarcoma (UPS), liposarcoma (LPS), leiomyosarcoma (LMS), synovial sarcoma ( SS). The most common soft tissue sarcoma in children and adolescents is rhabdomyosarcoma (RMS). Soft tissue sarcoma is a group of highly heterogeneous tumors, which are characterized by local invasiveness, invasive or destructive growth, local recurrence and distant metastasis.

The pathological features of STS that occur in the nasal cavity and sinuses are similar to other parts of the body. However, because it can affect important structures such as the orbit, optic nerve, skull base bone, dura mater, cranial nerve and even brain tissue, the diseased site is deep, the anatomical structure is complex, the treatment is difficult, the range of surgical resection is limited, and the surgical margin Negative is difficult to guarantee, and related treatments may have obvious complications, which affect the survival and prognosis of patients.

Surgical treatment is the most important and most likely effective treatment for STS. With the development of endoscopic skull base anatomy and surgical techniques, the safety and effectiveness of endoscopic sinus surgery for the treatment of nasal cavity and sinus tumors have been fully confirmed, and it has become the main surgical method for nasal cavity and sinus STS. This is also the theoretical and practical basis for the feasibility of this research.

The study intends to conduct a single-arm, prospective, observational study of endoscopic sinus surgery for the treatment of soft tissue sarcoma of the nasal cavity and paranasal sinuses to explore the therapeutic effect and complications of endoscopic surgery for the treatment of soft tissue sarcoma of the nasal cavity and paranasal sinuses, and explore its relationship with chemotherapy and radiotherapy. The model of comprehensive treatment between.

DETAILED DESCRIPTION:
The study intends to conduct a single-arm, prospective, observational study of endoscopic sinus surgery for the treatment of soft tissue sarcoma of the nasal cavity and paranasal sinuses to explore the therapeutic effect and complications of endoscopic surgery for the treatment of soft tissue sarcoma of the nasal cavity and paranasal sinuses, and explore its relationship with chemotherapy and radiotherapy. The model of comprehensive treatment between.This study is divided into a screening period, a treatment period, and a follow-up period. All subjects need to sign an informed consent form before screening, perform relevant blood tests, imaging examinations, and compare the inclusion and exclusion criteria to select suitable patients to enter the treatment period. The follow-up period is 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form;
2. STS of nasal cavity and paranasal sinuses diagnosed pathologically;
3. General physical condition can tolerate endoscopic sinus surgery;
4. There is no distant transfer;
5. The research team must believe that the patient can be completely removed by surgery;
6. Good organ function;

Exclusion Criteria:

1. The patient has surgical contraindications: such as severe cardiopulmonary disease, coagulation dysfunction;
2. Suffer from uncontrolled concurrent diseases;
3. There is a serious neurological or mental illness, including dementia and epileptic seizures;
4. Uncontrolled active infection;
5. There are any other circumstances that may hinder the compliance of the research;
6. Women who are pregnant or breastfeeding.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: For patients diagnosed with STS in the nasal cavity and paranasal sinuses through pathology, appropriate subjects will be selected according to the selection criteria and exclusion criteria of the protocol design.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-06-12 (Actual); Primary Completion 2023-06-12 (Estimated); Study Completion 2026-06-12 (Estimated)

PRIMARY OUTCOMES:
overall survival | From date of enrollment until the date of death from any cause, whichever came first，through study completion,up to 5 years.
  From the day of enrollment to death for any reason

SECONDARY OUTCOMES:
Local recurrence-free survival | From date of first treatment until the date of local recurrence or the date of death from any cause,through study completion,up to 5 years.
  The time from enrollment to local recurrence or death for any reason
quality of life | within 1 year after surgery
  The Chinese version of EORTC QLQ C30 questionnaire (V3.0)

CONTACTS AND LOCATIONS:
Locations (1):
- Yu Hongmeng, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
undecided